CLINICAL TRIAL: NCT04945343
Title: Long-Term Follow-Up Of Surgical Management Of Early Onset Scoliosis Using Growing Rods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Hatem Ahmed Mohammed, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Results of growing rods
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Early-Onset Scoliosis Deformity of Spine
Keywords: Growing rods; Scoliosis; Pediatric spine deformity
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Use of growing Rods for correction of early onset scoliosis deformity of the spine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children who had growing rods instrumentation for correction of Early Onset Scoliosis (Other): Growing spine profiler instrumentation
  Interventions: Procedure: Growing Rods

INTERVENTIONS:
Procedure: Growing Rods — Growing Rods(GR), are implants used to correct pediatric scoliosis deformity. They attempt to allow the growth of the spine and thorax while controlling curve progression to preserve normal lung volume.

SUMMARY:
The aim of this work is to evaluate the long-term outcome of the graduates (those who completed the gradual lengthening procedures), to better understand the full scope and natural course of Growing Rods treatment for EOS and to have a glimpse of what happens to the graduates.

DETAILED DESCRIPTION:
The management of progressive early onset scoliosis (EOS) is challenging. The natural history can be severe deformity, restrictive lung disease, and early mortality . In the past, the standard of care for these children was early definitive spinal fusion and instrumentation. The belief was that a short and straight spine was superior to a long and deformed spine despite the negative effects of a short trunk. The principles of EOS treatment have changed with the appreciation that early fusion of the thoracic spine limits the growth of the spine and lungs, and eventually leads to respiratory failure and increased mortality. Furthermore, the cosmetic disfigurement from the disproportionate Trunk-Limb length is always not acceptable by the patients.

The surgical treatment strategy for EOS has evolved significantly with the use of modern growth friendly implants, of these, Growing Rods(GR), first described by Moe and colleagues, attempt to allow the growth of the spine and thorax while controlling curve progression to preserve normal lung volume. Since then, several modifications and developments have been made and introduced worldwide.

Evaluation of the mid to long-term follow up has seldom been reported in the literature. In Assiut university hospital the investigators operated a fair amount of children with EOS using growing rods starting 2009, with favourable short term results. The long-term outcome of the graduates (those who completed the gradual lengthening procedures), remains yet to be evaluated and reported.

Research Methods and techniques:

Type of the study: case series

Study Setting: Assiut University Hospitals, Department of Orthopaedics, Spine Surgery Unit.

Study subjects:

1. Inclusion criteria:

   Any patient with EOS who has been managed with GRs in our centre.
2. Exclusion criteria:

   Patients whose parents or guardians are not willing to participate in the study.
3. Sample Size Calculation:

All patients with EOS operated in our centre who have completed the GR procedures and became graduates since we started doing surgeries in 2009 to the present date. We expect to have complete data for 30 patients during the study period.

-Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, ):

* Data sheet (Personal data, Cobb's angle, kyphosis angle, Shoulder balance, Coronal and sagittal balance, Pelvic obliquity, T1-S1 height,Span-Height ratio, patient satisfaction score (Likert scale).
* Early Onset Scoliosis 24-Item Questionnaire (EOSQ-24) Arabic version .
* Radiological assessment (Cobb's angle, kyphosis angle, Shoulder balance, Coronal and sagittal balance, Pelvic obliquity, T1-S1 height, Implant Failure.)
* All data will be collected and recorded using the REDCap to facilitate data recording, analysis and creation of safe dedicated database.

Research outcome measures:

1. Primary (main):

   Percentage of improvement in the functional outcome of these patients using the EOSQ-24, Arabic Version)
2. Secondary (subsidiary):

   1-Patient satisfaction (Likert scale). 2 Trunk Height Gain (T1-S1 height). 3-Span-Height ratio. 4-The degree of correction of the scoliosis and kyphosis. 5-Maintenance of sagittal and coronal balance. Incidence of complications (PJK, DJK, recurrent infections, neurology, crankshaft phenomenon, etc)

ELIGIBILITY:
Inclusion criteria:

-Any patient with EOS who has been managed with GRs in our centre.

Exclusion Criteria:

* Patients whose parents or guardians are not willing to participate in the study.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement in the functional outcome of these patients using the EOSQ-24, Arabic Version) | Through study completion, an average of 2 years.
  A score that measures the wider dimensions of outcomes involving the quality of life of patients and caregivers post-treatment.

SECONDARY OUTCOMES:
Patient satisfaction (Likert scale) | Through study completion, an average of 2 years.
  A five point scale which is used to allow the individual to express how much they are satisified or unsatisified with the outcomes.
Trunk Height Gain (T1-S1 height). | Through study completion, an average of 2 years.
  The vertical distance from the midpoint of the superior endplate of T1 to the midpoint of the superior endplate of S1.
The degree of correction of the scoliosis and kyphosis. | Through study completion, an average of 2 years.
  measured through Cobb's angle
sagittal and coronal balance | Through study completion, an average of 2 years.
  measured through the C7 plumb line and the central sacral vertical line respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad El-Sharkawi, professor, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals,department of Orthopaedics,Spine surgery unit., Asyut, Egypt